CLINICAL TRIAL: NCT03362814
Title: A Phase2/3, Multi-center, Randomized, Double-blind, Placebo-parallel Controlled Study to Investigate the Efficacy and Safety of Ravidasvir in Combination With Danoprevir/r and Ribavirin(RBV) in Treatment-naive, Non-cirrhotic, Chronic Hepatitis C Genotype 1 Infected Subjects.
Brief Title: Efficacy and Safety of Ravidasvir in Combination With Danoprevir/r and Ribavirin(RBV) in Treatment-naive, Non-cirrhotic, Chronic Hepatitis C Virus Genotype1 Infected Subjects.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC-ASC16-II/III-CTP-1-01
Record Dates: First submitted 2017-11-28; First posted 2017-12-05 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2017-11

CONDITIONS: HCV
Keywords: HCV; Ravidasvir; SVR12
MeSH Terms: interventions — ravidasvir; danoprevir; Ritonavir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Ravidasvir + Danoprevir + Ritonavir + Ribavirin
  Interventions: Drug: Ravidasvir; Drug: Danoprevir; Drug: Ritonavir; Drug: Ribavirin 100 MG
- Placebo Group (Placebo Comparator): Ravidasvir placebo + Danoprevir placebo + Ritonavir placebo + Ribavirin placebo
  Interventions: Drug: Ravidasvir Placebo; Drug: Danoprevir Placebo; Drug: Ritonavir Placebo; Drug: Ribavirin Placebo

INTERVENTIONS:
Drug: Ravidasvir — Ravidasvir 200mg tablet administered orally once daily
  Other Names: ASC16
  Arms: Experimental Group
Drug: Danoprevir — Danoprevir 100mg tablet administered orally twice daily
  Other Names: ASC08
  Arms: Experimental Group
Drug: Ritonavir — Ritonavir 100mg tablet administered orally twice daily
  Arms: Experimental Group
Drug: Ribavirin 100 MG — Ribavirin tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations(<75kg = 1000mg and ≥75kg = 1200mg)
  Arms: Experimental Group
Drug: Ravidasvir Placebo — Ravidasvir Placebo tablet administered orally once daily
  Arms: Placebo Group
Drug: Danoprevir Placebo — Danoprevir Placebo tablet administered orally twice daily
  Arms: Placebo Group
Drug: Ritonavir Placebo — Ritonavir Placebo tablet administered orally twice daily
  Arms: Placebo Group
Drug: Ribavirin Placebo — Ribavirin Placebo tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations(<75kg = 5 tablets and ≥75kg = 6 tablets)
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Ravidasvir in combination with Danoprevir/r and ribavirin(RBV) by sustain virologic response 12 (SVR12), in treatment-naive, non-cirrhotic, chronic hepatitis C genotype 1 infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Infection with Chronic hepatitis C genotype 1confirmed at screening;
* Anti-HCV positive；
* HCV RNA ≥1 × 10000IU / mL;
* Not treated with interferon and / or any other direct-acting antiviral (DAA) drug;
* Non-cirrhotic;
* Voluntarily sign informed consent.

Exclusion Criteria:

* HCV genotypes 2 to 7 or undetectable HCV genotype or mixed HCV genotype;
* Fibroscan detection result > 12.9kPa or Histopathological examination result of patients is with cirrhosis;
* Past or existing evidence of the presence of non-HCV-induced chronic liver disease;
* Previous history of hepatocellular carcinoma, or suspected hepatocellular carcinoma found prior to screening, or suspected abdominal hepatoblastoma at screening or AFP>100ng/mL;
* Anti-HAV (IgM) 、HBsAg 、anti-HEV (IgM) or anti-HIV is positive;
* BMI<18 or≥30 kg/m2;
* ANC<1.5×109/L、PLT<100×109/L、HB<110g/L（female）or<120g/L（male）；INR>1.5；ALT or AST≥5*ULN；TBIL≥2*ULN（DBIL≥ 35%TBIL）；Cr≥1.5*ULN;
* Others as specified in detailed protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants achieving sustained Virologic response 12 weeks after EOT | Post treatment Week 12
  SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) 12 weeks after cessation of therapy
Adverse events leading to permanent discontinuation of study drug | baseline to week 12

SECONDARY OUTCOMES:
Percentage of Participants achieving sustained Virologic response 4 weeks after EOT | Post treatment Week 4
  SVR4 was defined as HCV RNA < the lower limit of quantitation (LLOQ) 4 weeks after cessation of therapy
Percentage of Participants achieving sustained Virologic response 24 weeks after EOT | Post treatment Week 24
  SVR24 was defined as HCV RNA < the lower limit of quantitation (LLOQ) 24 weeks after cessation of therapy
Quatitation change of HCV RNA compared to baseline after treatment | Baseline to week 1
Percentage of participants with viral breakthrough | Baseline to week 12
  Viral breakthrough was defined as HCV RNA ≥LLOQ after having previously had HCV RNA< LLOQ while receiving treatment, confirmed with 2 consecutive values
Percentage of participants with viral relapse | End of treatment to post-treatment week 24
  Viral relapse was defined as HCV RNA ≥LLOQ during the post treatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values.

CONTACTS AND LOCATIONS:
Overall Officials: Yahong Chen, Master, Study Director — Ascletis Pharmaceuticals Co., Ltd.
Locations (1):
- Peking University People's hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No